CLINICAL TRIAL: NCT01044433
Title: A Phase II Study of Capecitabine and Lapatinib in Squamous Cell Carcinoma of the Head and Neck
Brief Title: Capecitabine and Lapatinib Ditosylate in Treating Patients With Squamous Cell Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 15309; NCI-2009-01492
Record Dates: First submitted 2009-12-10; First posted 2010-01-07 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer; Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral lapatinib ditosylate once daily on days 1-21 and oral capecitabine twice daily on days 1-14.
  Interventions: Drug: lapatinib ditosylate; Drug: capecitabine

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; lapatinib; Tykerb
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving capecitabine together with lapatinib ditosylate may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine and lapatinib ditosylate together works in treating patients with squamous cell cancer of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Overall survival (OS) will be the primary endpoint.

SECONDARY OBJECTIVES:

I. Progression free survival (PFS). II. Time to disease progression and sites of progression. III. Response rate. IV. Toxicity of the combination in this population. V. Quality of life.

OUTLINE:

Patients receive oral lapatinib ditosylate once daily on days 1-21 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion

* Histologically or cytologically confirmed SCCHN
* All primary sites are eligible excluding nasopharyngeal
* Metastatic disease or locally recurrent disease not felt amenable to curative therapy (as determined by a physician)
* ECOG performance status 0-2
* No prior chemotherapy in the metastatic / locally advanced, recurrent incurable setting; patients may have received prior curative-intention chemotherapy including induction chemotherapy, chemotherapy concurrent with radiation and adjuvant chemotherapy
* No prior capecitabine; patients who have received 5-FU or other fluoropyrimidines in the curative-intention setting will not be excluded, as long as more than 6 mos have elapsed since prior 5-FU exposure
* No previous history of Lapatinib
* Previous use of cetuximab in the curative-intention setting will not result in exclusion, as long as at least four weeks have elapsed since prior C225 exposure
* Patients may have received radiation therapy in the definitive, adjuvant or metastatic setting; radiation therapy must be completed at least 14 days prior to study participation
* ECOG performance status of 0-2 (Karnofsky >= 60%)
* Must have normal organ and marrow function
* Laboratory tests should be completed within 14 days prior to registration
* Left ventricular ejection fraction (LVEF) can be determined by either echocardiography or nuclear scintigraphy and should be obtained within 21 days of enrollment
* Platelets >= 100,000/mm^3
* Total bilirubin =< 2
* Albumin > 2.5
* AST(SGOT)/ALT(SGPT) =< 5.0 X institutional upper limit of normal (for patients with hepatic metastases) =< 3.0 X institutional upper limit of normal (for patients without hepatic metastases)
* GFR > 30 (by standard Cockroft and Gault formula)
* LVEF >= 50%
* Patients may receive anticoagulant medication while on study
* Patients may not receive other antineoplastic therapies such as chemotherapy or radiation treatments while on study; patients may not receive other experimental treatments while on study; patients requiring radiation treatments during protocol-based treatment will be taken off study
* Patients may receive concurrent bisphosphonate therapy as well as hormonal manipulations for appetite while on study
* Patients must neither be pregnant nor expect to become pregnant while on study
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Adequate swallowing function or gastric-tube for drug administration
* No disability with absorption of internal medications
* Adequate nutritional status: Patients will not be excluded based on previous weight loss but will be required to have adequate nutrition at the time of study entry as measured by serum albumin
* ANC >= 1,500/mm^3
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion

* Patients who have received prior capecitabine chemotherapy or lapatinib
* Patients with brain metastases may participate if they have undergone appropriate treatment for the lesion(s), are at least two weeks post treatment without evidence for post-treatment progression, have no significant neurologic symptoms, and are no longer on steroids for brain metastases
* Patients with symptoms concerning for CNS metastases should be evaluated with imaging prior to study participation
* Less than 3 weeks elapsed since prior exposure to chemotherapy
* LVEF < 50% or symptomatic congestive heart failure (CHF)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded due to the potential for teratogenic or abortifacient effects of capecitabine and lapatinib; because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued prior to participation of the mother on study
* Other active, invasive malignancy requiring ongoing therapy or expected to require systemic therapy within two years; localized squamous cell carcinoma of the skin, basal-cell carcinoma of the skin, carcinoma in-situ of the cervix, or other malignancies requiring locally ablative therapy only will not result in exclusion
* Have received treatment within the last 30 days prior to study entry with any drug that has not received regulatory approval for an indication at the time of study entry
* Previous CHF or other cardiac conditions shall not result in exclusion if the treating physician does not see contraindication to these medications; if contraindication is controversial, cardiac consultation will be obtained prior to the initiation of therapy
* Anti-cancer therapy (other than the investigational regimen) is prohibited from 3 weeks before the first dose of investigational product through discontinuation unless otherwise noted
* Investigational drugs are not permitted from 3 weeks (21 days) or 5 half-lives, whichever is longer, prior to the first dose and up through 30 days after the last dose of investigational product
* CYP3A4 inducers and inhibitors, antacids, and herbal or dietary supplements
* Concurrent radiation therapy and surgery for SCCHN is prohibited during therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2015-09-24 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib Ditosylate and Capecitabine: Patients receive oral lapatinib ditosylate once daily on days 1-21 and oral capecitabine twice daily on days 1-14.
  lapatinib ditosylate: Given orally
  capecitabine: Given orally
Period: Overall Study
Arm/Group | Lapatinib Ditosylate and Capecitabine
Started | 44
Completed | 38
Not Completed | 6
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib Ditosylate and Capecitabine
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 5 years
Measure: Mean (90% Confidence Interval); unit: Months
Arm/Group | Lapatinib Ditosylate and Capecitabine
Number analyzed (Participants) | 44
Months | 10.7 [8.7 to 12.9]

2. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 5 years
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Arm I
Number analyzed (Participants) | 44
percentage | 25 [15 to 38]

3. Secondary Outcome: Disease Control Rate
Time Frame: 5 years
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Arm I
Number analyzed (Participants) | 44
percentage | 68 [55 to 80]

4. Secondary Outcome: Progression-free Survival
Time Frame: 5 years
Measure: Number (90% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 44
months | 4.2 [3.6 to 5.1]

5. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: ADVERSE EVENTS (AE) AND SERIOUS ADVERSE EVENTS (SAE) Adverse Events (AEs) will use the descriptions and grading scales found in the NCI CTCAE v3.0
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 44
Participants
  Diarrhea | 31
  Rash | 31
  Pain | 26
  Fatigue | 23
  Infection | 19
  Nausea | 19
  Mucositis | 14
  Vomiting | 13
  Constipation | 10
  Hand-foot syndrome | 8
  Cough | 7
  Acute kidney injury | 6
  Dry skin | 6
  Anorexia | 6
  Dehydration | 5
  Edema of limb | 5
  Heartburn | 5
  Hyponatremia | 5
  Neuropathy | 5
  Neutropenia | 2
  Febrile | 1

ADVERSE EVENTS:
Arm/Group | Lapatinib Ditosylate and Capecitabine
Serious Adverse Events (participants affected / at risk) | 44/44
Other Adverse Events (participants affected / at risk) | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Ditosylate and Capecitabine (N=44)
Diarrhea (Gastrointestinal disorders) | 31
Rash (Endocrine disorders) | 31
Pain (General disorders) | 26
Fatigue (General disorders) | 23
Infection (Infections and infestations) | 19
Nausea (Gastrointestinal disorders) | 19
Mucositis (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 10
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Acute kidney injury (Renal and urinary disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 5
Edema of limb (Vascular disorders) | 5
Heartburn (Gastrointestinal disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Neuropathy (Nervous system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 5
Febrile (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No